CLINICAL TRIAL: NCT00333762
Title: Use of "Smart Wheelchairs" to Provide Independent Mobility to Visual and Mobility Impairments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B4065-X
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-10

CONDITIONS: Blindness; Spinal Cord Injury
Keywords: aging; blindness; wheelchairs; spinal cord injury
MeSH Terms: conditions — Blindness; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPAM and SWCS (Experimental): Smart Power Assistance Module (SPAM) Smart Wheelchair Component System (SWCS)
  Interventions: Device: Smart Power Assistance Module (SPAM); Device: Smart Wheelchair Component System (SWCS)

INTERVENTIONS:
Device: Smart Power Assistance Module (SPAM) — Experimental Power wheelchair utilized to traverse prescribed course
Device: Smart Wheelchair Component System (SWCS) — Experimental power wheelchair utilized to traverse prescribed course

SUMMARY:
The goal of this project is to evaluate the Smart Wheelchair Component System (SWCS) for power wheelchairs and the Smart Power Assistance Module (SPAM) for manual wheelchairs in realistic indoor environments with target users performing realistic tasks. We will combine group trials involving individuals who have a visual impairment (but do not have a mobility impairment) with several single-case studio involving individuals who have a visual and mobility impairment. Our long-term objective is to provide independent mobility to veterans with mobility and sensory impairments.

DETAILED DESCRIPTION:
There are currently very few mobility options for veterans who have a mobility impairment and visual impairment, and this population will grow as the number of older veteran's increases. The goal of this project is to evaluate the Smart Wheelchair Component System (SWCS) for power wheelchairs and the Smart Power Assistance Module (SPAM) for manual wheelchairs in realistic indoor environments with target users performing realistic tasks. We will combine group trials involving individuals who have a visual impairment (and may or may not have a mobility impairment) with several single-case studies involving individuals who have a visual and mobility impairment.

The key questions that will be addresses by the proposed research are:

Can smart wheelchair technology improve performance on realistic navigation tasks for individuals with visual and mobility impairments?

Will smart wheelchair technology increase the amount of independent travel by individuals with visual and mobility impairments?

Will using a smart wheelchair for an extended period of time diminish a person's ability to operate a "traditional" wheeled mobility aid?

ELIGIBILITY:
Inclusion Criteria:

* All participants will be completely blind
* Participants will be able to operate a power wheelchair with joystick control
* Participants will be able to push a manual wheelchair a minimum of 300 yards

Exclusion Criteria:

* Mobility impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Simpson, PhD, Principal Investigator — VAPHS
Locations (2):
- United States (2):
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

REFERENCES:
- See also: Click here for more information about this study: Use of "Smart Wheelchairs" to Provide Independent Mobility to Visual and Mobility Impairments — http://www.herl.pitt.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: SWCS and SPAM: Subjects traversed a prescribed route using electric powered wheelchairs
  Smart Wheelchair Component System (SWCS) :
  Smart Power Assistance Module (SPAM) :
Period: Overall Study
Arm/Group | Arm 1: SWCS and SPAM
Started | 4
Completed | 0
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1: SWCS and SPAM
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Trial Wheelchair Course
Description: Time to complete the course was recorded. The indoor course was set up in the research laboratory to include a straight path and 90 degree turns that included obstacles such as a cardboard box, a large orange cone, and a desk chair. The location of these obstacles were randomly placed in order to test whether or not the SPAM or SWCS was able to detect objects.
Time Frame: Two years
Population: No data was collected.
Arm/Group | Arm 1: SWCS and SPAM
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Arm 1: SWCS and SPAM
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Only four subjects actually tested the chair. It was decided to stop after these four subject tests because the chairs were clearly not viable for this population of persons who were totally blind, and thus there was no need for further testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes